CLINICAL TRIAL: NCT02698709
Title: Astigmatic Vector Analysis of Posterior Corneal Surface - a Comparison Among Healthy, Forme Fruste and Overt Keratoconus Corneas
Brief Title: Astigmatic Vector Analysis of Posterior Cornea - a Comparison Among Healthy, Forme Fruste and Overt Keratoconus Corneas
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giuliano de Oliveira Freitas, MD., MD, University of Sao Paulo
Other Study IDs: Clínica Oftalmológica HCFM/USP
Record Dates: First submitted 2016-02-24; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal Topography; Diagnosis; Keratomileusis, Laser In Situ
MeSH Terms: conditions — Keratoconus; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy corneas (C): Corneas of normal candidates to refractive surgery who did not develop any sign of corneal ectasia after laser in situ keratomileusis during a two year follow-up period were analyzed by an Scheimpflug-based tomographer. Vector astigmatism analysis of anterior and posterior corneal surfaces were studied in accordance to method proposed by Thibos.
  Interventions: Other: Analysis of anterior and posterior corneal surfaces
- Overt keratoconus (Kc): Whether both eyes manifested classic Kc-suggestive topographic features, such as corneal steepness higher than 47.20 diopters (D), superior-inferior asymmetry higher than 1.40 D and thinnest pachymetric reading lower than 500 micrometers. Such eyes were analyzed by an Scheimpflug-based tomographer. Vector astigmatism analysis of anterior and posterior corneal surfaces were studied in accordance to method proposed by Thibos.
  Interventions: Other: Analysis of anterior and posterior corneal surfaces
- Forme fruste keratoconus (FFKc): Whether only one eye manifested classic Kc-suggestive topographic features, such as corneal steepness higher than 47.20 diopters (D), superior-inferior asymmetry higher than 1.40 D and thinnest pachymetric reading lower than 500 micrometers, and the fellow eye seemed unaffected. Such unaffected eyes were analyzed by an Scheimpflug-based tomographer. Vector astigmatism analysis of anterior and posterior corneal surfaces were studied in accordance to method proposed by Thibos.
  Interventions: Other: Analysis of anterior and posterior corneal surfaces

INTERVENTIONS:
Other: Analysis of anterior and posterior corneal surfaces — Corneal data obtained from a Scheimpflug-based topographer were converted to astigmatic vectors in accordance to the method proposed by Thibos
  Other Names: Thibos' vectorial astigmatism analysis

SUMMARY:
The main purpose of this study is to determine new diagnostic criteria for an eye disease called keratoconus.

DETAILED DESCRIPTION:
Eyes of patients who distinctly present signs of keratoconus, for both eyes, at corneal tomography (an exam commonly used in such cases), and those who present such signs in only one eye were compared to eyes of unaffected patients. Several characteristics of anterior and posterior corneal astigmatism (special emphasis was given to the latter) were collectively assessed among all patients by a method referred to as vectorial analysis. Statistical tests were then performed, in an attempt to highlight differences among those three groups of patients and, eventually, define new diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

* Good-quality Scheimpflug scans (approved by the device in the ''Examination Quality Specification'').

Exclusion Criteria:

* Previous eye surgery or trauma, and any sort of corneal scarring that might interfere with keratometric data acquisition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two databases of patients were examined at the Instituto de Olhos Renato Ambrósio (Rio de Janeiro, Brazil), between July 2004 and October 2013. One of the databases contained information of normal candidates to refractive surgery who did not develop any sign of corneal ectasia after laser in situ keratomileusis during a two year follow-up period (C). The second database included information concerning corneas with keratoconus (Kc), categorized as overt Kc, if both eyes manifested classic Kc-suggestive topographic features, such as corneal steepness higher than 47.20 diopters (D), superior-inferior asymmetry higher than 1.40 D and thinnest pachymetric reading lower than 500 micrometers; or forme fruste (FFKc), if only one eye exhibited such features.
Sampling Method: Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Astigmatism corneal vectors (based on keratometric readings at the three millimeter optical zones for both corneal surfaces). | Through study completion, an average of 6 months.
  Corneal tomography at an Scheimpflug-based tomographer

CONTACTS AND LOCATIONS:
Overall Officials: Milton R Alves, MD, PhD, Study Director — Clínica Oftalmológica HCFM/USP
Locations (1):
- Clínica Oftalmológica do Hospital de Clínicas - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li X, Yang H, Rabinowitz YS. Keratoconus: classification scheme based on videokeratography and clinical signs. J Cataract Refract Surg. 2009 Sep;35(9):1597-603. doi: 10.1016/j.jcrs.2009.03.050. PMID 19683159
- [Result] Goebels S, Eppig T, Wagenpfeil S, Cayless A, Seitz B, Langenbucher A. Staging of keratoconus indices regarding tomography, topography, and biomechanical measurements. Am J Ophthalmol. 2015 Apr;159(4):733-8. doi: 10.1016/j.ajo.2015.01.014. Epub 2015 Jan 26. PMID 25634534
- [Result] Moreira LB, Bardal RA, Crisigiovanni LR. Contact lenses fitting after intracorneal ring segments implantation in keratoconus. Arq Bras Oftalmol. 2013 Jul-Aug;76(4):215-7. doi: 10.1590/s0004-27492013000400004. PMID 24061830
- [Result] Raiskup F, Theuring A, Pillunat LE, Spoerl E. Corneal collagen crosslinking with riboflavin and ultraviolet-A light in progressive keratoconus: ten-year results. J Cataract Refract Surg. 2015 Jan;41(1):41-6. doi: 10.1016/j.jcrs.2014.09.033. PMID 25532633
- [Result] Gomes JA, Tan D, Rapuano CJ, Belin MW, Ambrosio R Jr, Guell JL, Malecaze F, Nishida K, Sangwan VS; Group of Panelists for the Global Delphi Panel of Keratoconus and Ectatic Diseases. Global consensus on keratoconus and ectatic diseases. Cornea. 2015 Apr;34(4):359-69. doi: 10.1097/ICO.0000000000000408. PMID 25738235
- [Result] Muftuoglu O, Ayar O, Ozulken K, Ozyol E, Akinci A. Posterior corneal elevation and back difference corneal elevation in diagnosing forme fruste keratoconus in the fellow eyes of unilateral keratoconus patients. J Cataract Refract Surg. 2013 Sep;39(9):1348-57. doi: 10.1016/j.jcrs.2013.03.023. Epub 2013 Jun 29. PMID 23820305
- [Result] Smadja D, Santhiago MR, Mello GR, Krueger RR, Colin J, Touboul D. Influence of the reference surface shape for discriminating between normal corneas, subclinical keratoconus, and keratoconus. J Refract Surg. 2013 Apr;29(4):274-81. doi: 10.3928/1081597X-20130318-07. PMID 23557226
- [Result] Torricelli AA, Bechara SJ, Wilson SE. Screening of refractive surgery candidates for LASIK and PRK. Cornea. 2014 Oct;33(10):1051-5. doi: 10.1097/ICO.0000000000000171. PMID 25014146
- [Result] Randleman JB, Akhtar J, Lynn MJ, Ambrosio R Jr, Dupps WJ Jr, Krueger RR, Klyce SD. Comparison of objective and subjective refractive surgery screening parameters between regular and high-resolution Scheimpflug imaging devices. J Cataract Refract Surg. 2015 Feb;41(2):286-94. doi: 10.1016/j.jcrs.2014.06.026. Epub 2014 Dec 20. PMID 25537685
- [Result] Ramos IC, Correa R, Guerra FP, Trattler W, Belin MW, Klyce SD, Fontes BM, Schor P, Smolek MK, Dawson DG, Chalita MR, Cazal JO, Ruiz M, Randleman JB, Ambrosio R Jr. Variability of subjective classifications of corneal topography maps from LASIK candidates. J Refract Surg. 2013 Nov;29(11):770-5. doi: 10.3928/1081597X-20130823-01. Epub 2013 Aug 30. PMID 23980708
- [Result] Qin B, Chen S, Brass R, Li Y, Tang M, Zhang X, Wang X, Wang Q, Huang D. Keratoconus diagnosis with optical coherence tomography-based pachymetric scoring system. J Cataract Refract Surg. 2013 Dec;39(12):1864-71. doi: 10.1016/j.jcrs.2013.05.048. PMID 24427794
- [Result] Ruisenor Vazquez PR, Galletti JD, Minguez N, Delrivo M, Fuentes Bonthoux F, Pfortner T, Galletti JG. Pentacam Scheimpflug tomography findings in topographically normal patients and subclinical keratoconus cases. Am J Ophthalmol. 2014 Jul;158(1):32-40.e2. doi: 10.1016/j.ajo.2014.03.018. Epub 2014 Apr 5. PMID 24709808
- [Result] Buhren J, Schaffeler T, Kohnen T. Validation of metrics for the detection of subclinical keratoconus in a new patient collective. J Cataract Refract Surg. 2014 Feb;40(2):259-68. doi: 10.1016/j.jcrs.2013.07.044. Epub 2013 Dec 18. PMID 24360499
- [Result] Galletti JD, Ruisenor Vazquez PR, Minguez N, Delrivo M, Bonthoux FF, Pfortner T, Galletti JG. Corneal asymmetry analysis by pentacam scheimpflug tomography for keratoconus diagnosis. J Refract Surg. 2015 Feb;31(2):116-23. doi: 10.3928/1081597X-20150122-07. PMID 25735045
- [Result] Ambrosio R Jr, Valbon BF, Faria-Correia F, Ramos I, Luz A. Scheimpflug imaging for laser refractive surgery. Curr Opin Ophthalmol. 2013 Jul;24(4):310-20. doi: 10.1097/ICU.0b013e3283622a94. PMID 23680761
- [Result] Montalban R, Pinero DP, Javaloy J, Alio JL. Scheimpflug photography-based clinical characterization of the correlation of the corneal shape between the anterior and posterior corneal surfaces in the normal human eye. J Cataract Refract Surg. 2012 Nov;38(11):1925-33. doi: 10.1016/j.jcrs.2012.06.050. Epub 2012 Sep 14. PMID 22981614
- [Result] Montalban R, Pinero DP, Javaloy J, Alio JL. Correlation of the corneal toricity between anterior and posterior corneal surfaces in the normal human eye. Cornea. 2013 Jun;32(6):791-8. doi: 10.1097/ICO.0b013e31827bf898. PMID 23328698
- [Result] Koch DD, Ali SF, Weikert MP, Shirayama M, Jenkins R, Wang L. Contribution of posterior corneal astigmatism to total corneal astigmatism. J Cataract Refract Surg. 2012 Dec;38(12):2080-7. doi: 10.1016/j.jcrs.2012.08.036. Epub 2012 Oct 12. PMID 23069271
- [Result] Pinero DP, Alio JL, Tomas J, Maldonado MJ, Teus MA, Barraquer RI. Vector analysis of evolutive corneal astigmatic changes in keratoconus. Invest Ophthalmol Vis Sci. 2011 Jun 8;52(7):4054-62. doi: 10.1167/iovs.10-6856. PMID 21372010
- [Result] Saad A, Gatinel D. Topographic and tomographic properties of forme fruste keratoconus corneas. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5546-55. doi: 10.1167/iovs.10-5369. Epub 2010 Jun 16. PMID 20554609
- [Result] Thibos LN, Horner D. Power vector analysis of the optical outcome of refractive surgery. J Cataract Refract Surg. 2001 Jan;27(1):80-5. doi: 10.1016/s0886-3350(00)00797-5. PMID 11165859
- [Result] Read SA, Collins MJ. Diurnal variation of corneal shape and thickness. Optom Vis Sci. 2009 Mar;86(3):170-80. doi: 10.1097/OPX.0b013e3181981b7e. PMID 19182699
- [Result] Eom Y, Rhim JW, Kang SY, Kim SW, Song JS, Kim HM. Toric Intraocular Lens Calculations Using Ratio of Anterior to Posterior Corneal Cylinder Power. Am J Ophthalmol. 2015 Oct;160(4):717-24.e2. doi: 10.1016/j.ajo.2015.07.011. Epub 2015 Jul 26. PMID 26215437
- [Result] Alpins N, Ong JK, Stamatelatos G. Corneal topographic astigmatism (CorT) to quantify total corneal astigmatism. J Refract Surg. 2015 Mar;31(3):182-6. doi: 10.3928/1081597X-20150224-02. PMID 25751835
- [Result] Gilani F, Cortese M, Ambrosio RR Jr, Lopes B, Ramos I, Harvey EM, Belin MW. Comprehensive anterior segment normal values generated by rotating Scheimpflug tomography. J Cataract Refract Surg. 2013 Nov;39(11):1707-12. doi: 10.1016/j.jcrs.2013.05.042. Epub 2013 Sep 18. PMID 24054966
- [Result] Lopes B, Ramos I, Ambrosio R Jr. Corneal densitometry in keratoconus. Cornea. 2014 Dec;33(12):1282-6. doi: 10.1097/ICO.0000000000000266. PMID 25285589
- [Result] Baratloo A, Hosseini M, Negida A, El Ashal G. Part 1: Simple Definition and Calculation of Accuracy, Sensitivity and Specificity. Emerg (Tehran). 2015 Spring;3(2):48-9. No abstract available. PMID 26495380
- [Result] Saunders LJ, Zhu H, Bunce C, Dore CJ, Freemantle N, Crabb DP; Ophthalmic Statistics Group. Ophthalmic statistics note 5: diagnostic tests-sensitivity and specificity. Br J Ophthalmol. 2015 Sep;99(9):1168-70. doi: 10.1136/bjophthalmol-2014-306055. Epub 2014 Dec 8. PMID 25488948
- [Result] McGee S. Simplifying likelihood ratios. J Gen Intern Med. 2002 Aug;17(8):646-9. doi: 10.1046/j.1525-1497.2002.10750.x. PMID 12213147
- [Result] Shi R, Conrad SA. Correlation and regression analysis. Ann Allergy Asthma Immunol. 2009 Oct;103(4 Suppl 1):S35-41. doi: 10.1016/s1081-1206(10)60820-4. No abstract available. PMID 19891286